CLINICAL TRIAL: NCT05496452
Title: Effect of Beta-lactoglobulin Supplementation on the Response of Muscle Protein Synthesis During Limb Immobilisation in Healthy Young Adults
Brief Title: Beta-lactoglobulin, Immobilisation and Muscle Protein Synthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BLGIMMPS
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2022-08

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — Lactoglobulins; Carbohydrates

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, 2-arm, randomised placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Double blinded to supplement (beta-lactoglobulin or carbohydrate)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-lactoglobulin (Experimental): Daily supplementation over 12 day period. A nutritional supplement.
  Interventions: Dietary Supplement: Beta-lactoglobulin
- Carbohydrate (Placebo Comparator): Daily supplementation over 12 day period. Energy matched control.
  Interventions: Dietary Supplement: Carbohydrate

INTERVENTIONS:
Dietary Supplement: Beta-lactoglobulin — Beta-lactoglobulin (BLG) will be administered thrice daily during a 7 day period of prehabilitation and 5 day period of immobilisation when the leg is placed in a brace.
  Arms: Beta-lactoglobulin
Dietary Supplement: Carbohydrate — Carbohydrate (dextrose monohydrate) will be administered thrice daily during a 7 day period of prehabilitation and 5 day period of immobilisation when the leg is placed in a brace.
  Arms: Carbohydrate

SUMMARY:
The objectives of this study are to:

1. Establish whether combined β-lactoglobulin supplementation and resistance training for 1 week prior to 5 days of limb immobilisation will attenuate the decrease in integrated free-living rates of MPS during short-term muscle disuse.
2. Establish whether combined β-lactoglobulin supplementation and resistance training for 1 week prior to limb immobilisation will attenuate the decrease in muscle mass and strength during short-term muscle disuse.

DETAILED DESCRIPTION:
The objectives of this study are to:

1. Establish whether combined β-lactoglobulin supplementation and resistance training for 1 week prior to 5 days of limb immobilisation will attenuate the decrease in integrated free-living rates of MPS during short-term muscle disuse.
2. Establish whether combined β-lactoglobulin supplementation and resistance training for 1 week prior to limb immobilisation will attenuate the decrease in muscle mass and strength during short-term muscle disuse.

Hypotheses

1. Combining β-lactoglobulin and resistance training for 1 wk prior to 5 d of limb immobilisation will attenuate the decrease in integrated muscle protein synthesis, muscle fibre CSA, quadriceps muscle strength, and leg lean mass during muscle disuse.
2. Combining β-lactoglobulin and resistance training for 1 wk prior to 5 d of limb immobilisation will attenuate the decrease in muscle fibre CSA, quadriceps muscle strength, and leg lean mass during muscle disuse.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Aged 18-45 years
* Healthy
* Physically active (≥150-300 minutes of moderate-intensity aerobic physical activity per week OR 75-150 minutes of vigorous-intensity aerobic physical activity per week)
* Eumenorrheic and not taking any hormonal birth control (females)

Exclusion Criteria:

* Dairy allergy or intolerance
* Lower limb injury or surgery in the last 6 months,
* Lower limb osteoarthritis or other musculoskeletal disorder
* A musculoskeletal or blood blotting disorder
* An allergy to local anaesthetic
* Currently pregnant
* Current use of blood thinning medications
* Volunteers that take part in structured resistance exercise training
* Taking supplements considered to be anabolic to skeletal muscle (protein supplements, creatine, or omega-3 supplements)
* Consuming more than 1.2 grams of protein per kilogram of body mass per day in their habitual diet.
* Volunteers involved in other studies at the time of enrolment
* Volunteers who have taken part in a tracer study in the past 18 months
* If without an understanding of verbal or written English
* Volunteers with a history of eating disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis | 15 days
  The synthesis of amino acids into new muscle protein.

SECONDARY OUTCOMES:
Muscle mass | 15 days
  Lean body mass will be measured using Dual Energy Xray Absorptiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Witard, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be presented in form of peer reviewed manuscript. While individual data will be presented, these data will not be identifiable to other researchers.

REFERENCES:
- [Derived] Hughes A, Francis T, Marjoram L, Rooney JH, Ellison-Hughes G, Pollock R, Curtis MJ, Cape A, Larsen M, Phillips BE, Atherton PJ, Smith K, Witard OC. The effect of combined beta-lactoglobulin supplementation and resistance exercise training prior to limb immobilisation on muscle protein synthesis rates in healthy young adults: study protocol for a randomised controlled trial. Trials. 2023 Jun 13;24(1):401. doi: 10.1186/s13063-023-07329-6. PMID 37312095